CLINICAL TRIAL: NCT01117597
Title: Experimental Study on Possible Effects of Radiofrequency (RF) Signal Characteristics Used for the TETRA Standard on Cognitive Functions in Healthy Subjects
Brief Title: Terrestrial Trunked Radio (TETRA) and Cognitive Functions in Healthy Subjects
Acronym: TETRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: The Federal Office for Radiation Protection, Germany (Other Government); Seibersdorf Labor GmbH (Industry)
Responsible Party: Principal Investigator, Heidi Danker-Hopfe, Prof. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: AVD20090991
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
Keywords: Healthy subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- low RF exposure level (Active Comparator): Intervention with low RF exposure level SAR 1.5 W/kg
  Interventions: Radiation: low RF exposure level
- sham RF exposure (Sham Comparator): Intervention with sham RF exposure
  Interventions: Radiation: sham exposure
- high RF exposure level (Active Comparator): intervention with high RF exposure level SAR 6W/kg
  Interventions: Radiation: high RF exposure

INTERVENTIONS:
Radiation: low RF exposure level — Exposure with 1.5 W/kg
  Arms: low RF exposure level
Radiation: sham exposure — intervention with sham RF exposure
  Arms: sham RF exposure
Radiation: high RF exposure — intervention with high RF exposure
  Arms: high RF exposure level

SUMMARY:
The purpose of this study is to analyse a possible effect of radiofrequency (RF) fields used for Terrestrial Trunked Radio (TETRA) of brain activity and cognitive functions in occupationally exposed subjects.

DETAILED DESCRIPTION:
Background

Several international studies on the influence of electromagnetic fields from mobile communications on cognitive performance and brain function during waking and sleep were performed during the last years. No health relevant effects were found below the maximum exposure of 2 Watt per kilogram (W/kg), which applies for the use of mobile devices by the public.

In Germany a new digital radio communication network for security authorities and organisations based on the TETRA standard is set up at present. TETRA (Terrestrial Trunked Radio) uses a frequency band around 400 MHz and has been much less investigated than public mobile communications. The results of the German Mobile Telecommunication Research Programme showed a higher temperature increase of the exposed tissue at 400 MHz than at the frequencies used by mobile phones. For occupational groups using mobile TETRA devices (as for example policemen and firemen), a local exposure up to 10 W/kg is permitted. Possible effects of electromagnetic fields of mobile TETRA devices will be investigated in humans to further reduce scientific uncertainties concerning the impact of the digital radio for security authorities.

Objective

In the present study, possible effects of an exposure with TETRA signals (sham, SAR values of 1.5 W/kg and 6 W/kg) on the brain activity of humans are investigated. A volunteer study is performed on healthy young men, preferentially from the group of potential users who will be occupationally exposed.

Tests are performed allowing conclusions on reaction speed and accuracy, processing of acoustic and visual information, ability to concentrate, memory and resilience.

In parallel, the waking EEG (electroencephalogram, examination of brain activity) under different conditions (rest, processing of tests) is recorded and evaluated.

Furthermore, the influence of TETRA exposure on sleep quality and sleep EEG, as well as performance and well being on the following day are investigated.

The results will be evaluated in relation to their health relevance for occupationally exposed users.

Volunteers

For study participation, young male subjects professionally engaged with TETRA at the age of 18 - 30 years are recruited, who are preferentially not active in night service, right handed and non-smokers.

1. Scientific knowledge

   In other European countries, security authorities have been using TETRA radio networks for some time. Similar to Germany, other European countries are actually setting up their nationwide networks. Some of these countries have accompanied the introduction of the TETRA standard by scientific research. At the beginning of the present study, the scientists of Charité Berlin performed a literature review on health effects of the digital radio bringing together data from publications and reports on the various national scientific results.

   Overall there are much less data for TETRA than for mobile communications. The few results published previously do not prove any health effects of TETRA.In one study a slight influence on memory was found, which could be by chance a result of the large amount of tests performed. Therefore this result has to be verified.

   Literature study (PDF, in German, 398 kB, not barrier-free)
2. Exposure setup

   In this study, volunteers are exposed in the head region to a TETRA signal at SAR values of 1.5 Watt per kilogram and 6 Watt per kilogram. A corresponding exposure setup was constructed and characterised by IMST GmbH (Kamp Lintfort). It is a flat antenna worn on the left side of the head which should simulate as far as possible exposures to a TETRA mobile device. It can be worn comfortably for up to eight hours, even during sleep. The true exposure of the individual brain regions was calculated in detail by Seibersdorf Laboratories GmbH.

   Description of the exposure setup (PDF, in German, 1,7 MB, not barrier-free)
3. Perception of warming

An exposure at SAR values of 6 W/kg causes a temperature increase in the head region of almost 1 ° C when using the exposure setup described above. Since the study is to be performed in a blinded way (neither the volunteer nor the directly involved scientist know the actual exposure situation) it is important to prove if the volunteers are able to perceive this warming. Therefore a pilot study was performed. It could be shown, that the volunteers are not able to recognize the actual temperature increase. Therefore, there is no risk of unblinding (the volunteers are not able to discover the specific exposure situation).

Report of the pilot study (PDF, 1,7 MB, in German, not barrier-free)

ELIGIBILITY:
Inclusion Criteria:

* healthy male subjects
* right handed
* potential TETRA users
* alpha-EEG
* non-smokers

Exclusion Criteria:

* acute illness
* severe neurological, psychiatric or internal disease
* ZNS-active medication
* sleep disorders
* drug abuse

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-04; Primary Completion 2013-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Performance in cognitive tests | acute effect under exposure will be assessed for a period of 3 hours for 9 test sessions (two weeks apart, three sessions for every exposure condition)

SECONDARY OUTCOMES:
Sleep quality | acute effect under exposure will be assessed for a period of approximately 8 hours for 9 experimental nights (two weeks apart, three nights for every exposure condition)

CONTACTS AND LOCATIONS:
Overall Officials: Blanka Pophof, PhD, Study Director — The Federal Office for Radiation Protection; Heidi Danker-Hopfe, PhD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Competence Sleep Medicine CC15, Charité University Medicine Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided